CLINICAL TRIAL: NCT06289322
Title: AI4HOPE - Artificial Intelligence Based Health, Optimism, Purpose and Endurance in Palliative Care for Dementia: Pilot Study 1 Digital Toolkit Assessment
Brief Title: AI4HOPE Pilot Study 1 Digital Toolkit Assessment
Acronym: AI4HOPE1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: University College Cork (Other); University of Leeds (Other); Fundacion Intras (Unknown); Universidade do Porto (Other); University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Lukas Radbruch, Director Department of Palliative Medicine, University Hospital Bonn, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EU101136769-CLIN1
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Toolkit for assessment of pain and distress (Other): A digital toolkit will be developed using facial emotional recognition and other instruments as well as questionnaires for the assessment of pain and distress in patients with dementia.
  Interventions: Other: Digital toolkit for assessment

INTERVENTIONS:
Other: Digital toolkit for assessment — The pilot study uses a digital assessment and intervention toolkit. The person with dementia and caregivers may choose from the digital interventions offered in the toolbox without any mandatory conditions.

SUMMARY:
The pilot study will develop and test a standardized assessment toolkit that will provide conclusive information with a tolerable burden for cognitively impaired patients with dementia.

DETAILED DESCRIPTION:
The clinical study is part of an EU-funded project on the use of artificial intelligence for patients with dementia. This study will test a digital toolkit fo assessment and monitoring of patients with mild or moderate dementia and pilot-test this toolkit for feasibility and acceptability.

Patients with mild to moderate dementia will be recruited for the pilot study in the six participating countries. The study population includes all types of dementia without stratification, as the aim of the study is to construct a digital assessment and intervention toolkit for clinical practice in any patient with cognitive impairment from any type of dementia.

Even though the final assessment and intervention toolkit could also be useful for patients with advanced dementia and more severe cognitive impairment, the pilot study will recruit only patients with mild or moderate dementia, who will still be able to provide informed consent, and who will be able to self-assess at least minimum patient-related outcome or patient-related experience measures to validate the behavioural and observational scales and biomarkers used in the toolkit.

Patients with dementia treated in the participating study centers will be screened for inclusion criteria and, if suitable will be invited to participate. The study will be performed for seven days, with optional extension to 30 days according to patients' preferences.

Patients with baseline data and at least one intervention performed from the digital toolkit and data completed before and after that intervention will be included in the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate dementia of any type
* Montrea Cognitive Assessment (MoCA) score of 16-25
* Living at home, or in residential or nursing home care
* Receiving adequate social support

Exclusion Criteria:

* Moderate/severe cognitive impairment (MoCA < 16)
* No cognitive impairment (MoCA >25)
* Inpatient or acute hospital treatment
* Infectious diseases or lokal skin conditons preventing the use of wearable body sensors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of toolkit | 7 days
  Patient feedback on feasibility, usefulness and burden of toolkit
Accuracy of toolkit assessments | 7 days
  Comparison of toolkit assessments of pain and distress (including facial emotional recognition from weekly diary recordings) and PROM/PREM.

SECONDARY OUTCOMES:
Effect of pain/distress interventions | 7 days
  Comparison of before/after assessments of interventions to alleviate pain or distress using the digital toolkit.
Exploration of specific linguistics and behavioural markers | Baseline, once per intervention week (at the end of the week)
  Exploration of specific linguistics and behavioural markers and their correlation with clinical assess-ment tools' scores.
Technology usability and usage metrics | At the end of intervention
  PROM/PREM completion rates, user engagement patterns, and dropout analysis.
Feedback on the diary interface | At the end of intervention
  Feedback on the diary interface and user experience that could inform future iterations.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Radbruch, MD, Principal Investigator — Department of Palliative Medicine, University Hospital Bonn

IPD SHARING:
Plan to Share IPD: No